# **Informed Consent Form (English Translation)**

Document Title: Informed Consent Form (English Translation)

Official Study Title: An Exploratory Study on the Dynamics of Dysbiosis in the Skin and Gut

Microbiome of Burn Patients

IRB Approval Number: HG2025-023 Document Date: September 8, 2025

Institution: Burn Institute, Hallym University Hangang Sacred Heart Hospital

Language: English Translation

#### 1. Basic Information

**Study Title:** An Exploratory Study on the Dynamics of Dysbiosis in the Skin and Gut Microbiome of Burn Patients

**Principal Investigator:** Prof. Yoon Soo Cho, Department of Rehabilitation Medicine, Hallym University Hangang Sacred Heart Hospital, Seoul, Republic of Korea.

This is a prospective observational study conducted in hospitalized burn patients to evaluate longitudinal changes in the skin and gut microbiome after burn injury.

#### 2. Study Description

This study aims to characterize the temporal dynamics of the skin and gut microbiome in burn patients, and understand dysbiosis and recovery patterns. Findings may inform future microbiome-based therapeutic strategies.

Participants: Adults (≥18 years) admitted for burn injuries.

Samples: Skin swabs (burned and non-burned), stool, and blood. Physiological skin parameters (TEWL, hydration, erythema, elasticity, pH) will be measured.

#### 3. Risks and Benefits

Risks: Minimal, such as mild skin irritation or redness. Benefits: No direct benefit, but may improve understanding of burn-related microbiome changes.

### 4. Costs and Compensation

There is no cost to participants and no financial compensation. Medical treatment will be provided at no cost for any study-related discomfort.

## 5. Voluntary Participation

Participation is voluntary, and withdrawal is allowed anytime without affecting medical care.

# 6. Confidentiality

All data will be de-identified and securely stored. Participant privacy will be maintained according to ethical standards.

### 7. Contact Information

Principal Investigator: Prof. Yoon Soo Cho

Tel: +82-2-2639-5730

Email: yschorm@hallym.ac.kr IRB Office: +82-2-2639-5900

## **Participant Consent**

I have read and understood the information above. I voluntarily agree to participate in this study. Participant's Name / Signature / Date Research Staff Name / Signature / Date Principal Investigator Signature / Date